CLINICAL TRIAL: NCT03691935
Title: Erector Spinae Plane Block (ESPB): A New Technique for Perioperative Pain Control in Patients Undergoing Surgery Through a Flank or Anterior Subcostal Incision.
Brief Title: Erector Spinae Plane Block (ESPB): in Patients Undergoing Surgery Through a Flank or Anterior Subcostal Incision.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment related to global pandemic and changes to surgical practice.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Alireza Aminsharifi, Assistant Professor of Surgery, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00008663
Record Dates: First submitted 2018-03-28; First posted 2018-10-02 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Nephrectomy; Partial Nephrectomy; Incision Site Discomfort
Keywords: kidney; surgery; analgesia; surgical incision; opioid sparing; flank pain; local anesthesia
MeSH Terms: conditions — Agnosia; Surgical Wound; Flank Pain | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivicaine (Experimental): Erector Spinae Block of 20ml 0.5% ropivicaine bolus, connected to a pump containing 0.2% ropivicaine receiving 15ml every 3 hrs.
  Interventions: Drug: Ropivacaine
- Normal Saline (Sham Comparator): Erector Spinae Block of 20ml normal saline placebo bolus, then connected to pump of normal saline receiving 15ml every 3 hrs.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ropivacaine — Erector Spinae Block with ropivacaine infusion with standard of care analgesics for perioperative pain control
  Other Names: Naropin
  Arms: Ropivicaine
Drug: Normal saline — Erector Spinae Block with saline infusion with standard of care analgesics for for perioperative pain control
  Other Names: Sham anesthetic
  Arms: Normal Saline

SUMMARY:
Using a randomized double-blinded study design, the study goal is to evaluate the superiority of Erector Spinae Plane block (ESPB) in the peri-operative pain management of patients undergoing surgery through a flank or anterior subcostal incision as compared to the standard of care of using IV and oral opiates.

DETAILED DESCRIPTION:
40 subjects will be randomized in to 2 groups, with 20 in each group.

* Group 1. Erector spinae plane block (ESPB) (containing Ropivacaine)
* Group 2. Sham Erector spinae plane block. (SESPB) (with normal saline)

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults age 18-85
* American Society of Anesthesiologists (ASA) Physical Status classification I to III
* Planned to be hospitalized for at least 24 hours post-op
* Cognitive capacity to use the visual analogic scale (VAS) and complete the patient satisfaction survey

Exclusion Criteria:

* Patient refusal
* Patients with allergies to local anesthetics or opiates (hydromorphone or oxycodone)
* Scoliosis
* Patients with chronic pain syndromes or who are on chronic pain medications/other neurologic medication of more than 3 months or whom have neuromodulators/stimulators
* Concurrent surgeries requiring additional incisions on the body

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Aminsharifi, M.D., Principal Investigator — Milton S. Hershey Medical Center; Sanjib Adhikary, M.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma V, Margreiter M. Partial nephrectomy: is there still a need for open surgery? Curr Urol Rep. 2013 Feb;14(1):1-4. doi: 10.1007/s11934-012-0297-2. PMID 23233109
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Gerbershagen HJ, Pogatzki-Zahn E, Aduckathil S, Peelen LM, Kappen TH, van Wijck AJ, Kalkman CJ, Meissner W. Procedure-specific risk factor analysis for the development of severe postoperative pain. Anesthesiology. 2014 May;120(5):1237-45. doi: 10.1097/ALN.0000000000000108. PMID 24356102
- [Background] de Beer Jde V, Winemaker MJ, Donnelly GA, Miceli PC, Reiz JL, Harsanyi Z, Payne LW, Darke AC. Efficacy and safety of controlled-release oxycodone and standard therapies for postoperative pain after knee or hip replacement. Can J Surg. 2005 Aug;48(4):277-83. PMID 16149361
- [Background] Recart A, Duchene D, White PF, Thomas T, Johnson DB, Cadeddu JA. Efficacy and safety of fast-track recovery strategy for patients undergoing laparoscopic nephrectomy. J Endourol. 2005 Dec;19(10):1165-9. doi: 10.1089/end.2005.19.1165. PMID 16359206
- [Background] Watcha MF, Issioui T, Klein KW, White PF. Costs and effectiveness of rofecoxib, celecoxib, and acetaminophen for preventing pain after ambulatory otolaryngologic surgery. Anesth Analg. 2003 Apr;96(4):987-994. doi: 10.1213/01.ANE.0000053255.93270.31. PMID 12651647
- [Background] Yenidunya O, Bircan HY, Altun D, Caymaz I, Demirag A, Turkoz A. Anesthesia management with ultrasound-guided thoracic paravertebral block for donor nephrectomy: A prospective randomized study. J Clin Anesth. 2017 Feb;37:1-6. doi: 10.1016/j.jclinane.2016.10.038. Epub 2016 Dec 15. PMID 28235492
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Continuous Erector Spinae Plane Block for Rescue Analgesia in Thoracotomy After Epidural Failure: A Case Report. A A Case Rep. 2017 May 15;8(10):254-256. doi: 10.1213/XAA.0000000000000478. PMID 28252539
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Gordon DB, Polomano RC, Pellino TA, Turk DC, McCracken LM, Sherwood G, Paice JA, Wallace MS, Strassels SA, Farrar JT. Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) for quality improvement of pain management in hospitalized adults: preliminary psychometric evaluation. J Pain. 2010 Nov;11(11):1172-86. doi: 10.1016/j.jpain.2010.02.012. Epub 2010 Apr 18. PMID 20400379

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivicaine | Normal Saline
Started | 11 | 9
Completed | 6 | 8
Not Completed | 5 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivicaine | Normal Saline | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13) | 61 (9.2) | 59 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores Using the Visual Analogue Pain Scale From Zero Pain to Level Ten Pain
Description: Data will be collected via the electronic medical record and begin following patient randomization. The Visual Analogue Scale pain scales will be administered and collected on Post Operative Days 1, 2 and 3. Minimum value = 0 No Pain, Maximum value = 10 Worst possible, unbearable, excruciating pain
Time Frame: Aggregate pain scores for average length of hospital stay which is 3 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropivicaine | Normal Saline
Number analyzed (Participants) | 6 | 8
units on a scale | 3.55 (1.2) | 4.6 (2.15)

ADVERSE EVENTS:
Time Frame: From enrollment to 14 days post-op for each subject
Arm/Group | Ropivicaine | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/9
Other Adverse Events (participants affected / at risk) | 3/11 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ropivicaine (N=11) | Normal Saline (N=9)
Post-op ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ropivicaine (N=11) | Normal Saline (N=9)
Increased pain (General disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed due Covid-19 and changes to surgical practice standard of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT03691935/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT03691935/ICF_001.pdf